CLINICAL TRIAL: NCT01537926
Title: Pilot Feasibility Study With N-acetylcystein (NAC) in Patients With HCM Caused by Sarcomere Proteins Mutations
Brief Title: Hypertrophic Regression With N-Acetylcysteine in HCM
Acronym: HALT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ali. J. Marian, Professor , Cardiovascular Genetics, IMM, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HALT-HCM; IR34HL105563 (Other: NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: HALT; HCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (NAC) (Experimental): N-acetylcysteine 600mg by mouth every 12 hours for 90 days. N-acetylcysteine 1200mg by mouth every 12 hours for 270 days
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Placebo 1 cap by mouth every 12 hours for 90 days. Placebo 2 caps by mouth every 12 hours for 270 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — NAC 600mg capsule or matching Placebo , 1 twice daily for 90 days, then increase to NAC 1,200mg or matching placebo, 2 capsules twice daily for 270 days.
  Other Names: NAC
  Arms: N-acetylcysteine (NAC)
Drug: Placebo — sugar pill manufactured to minic NAC 600mg capsule
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of the sudy is to conduct a small study to gather the preliminary data for future lage scale clinical studies that will be designed test the potential beneficial effect of over-the counter study anti-oxidant drug called N-acetylcysteine (NAC) in patients with a heart muscle condition called Hypertrophic Cardiomyopathy (HCM). The present study is a pilot feasibility study, the investigators want to find out whether the investigators can recruit and retain patients with HCM in the study and whether these patients can tolerate this drug and can stay on one year. Likewise, the investigators want to find out any potential side effects that this drug might have and estimate whether it has any beneficial effects.

DETAILED DESCRIPTION:
The primary objective is to perform a pilot study in patients with hypertrophic cardiomyopathy (HCM) and mutations in genes encoding sarcomere proteins to assess safety and gather the pre-requisite data for subsequent robust randomized placebo-controlled efficacy studies with N-acetylcysteine (NAC). Data will be gathered on the recruitment, accrual, retention, and compliance rates of HCM patients randomized to treatment with a placebo or two escalating doses of NAC. Likewise, any potential side effects will be determined and the effect size of NAC on indices of cardiac hypertrophy will be estimated. HCM, the main focus of the study team's research during the past two decades, is the most common cause of sudden cardiac death (SCD) in the young and an important cause of morbidity in the elderly. Despite its clinical impact, there is no effective pharmacological therapy for HCM. None of the current pharmacological therapies reverses or attenuates cardiac hypertrophy or reduces the risk of SCD in adults. Cardiac hypertrophy, the quintessential clinical feature of human HCM, is a major determinant of morbidity and the risk of SCD. Regression of cardiac hypertrophy is expected to improve morbidity and decrease the risk of SCD in HCM, as observed upon regression of load-dependent cardiac hypertrophy. The study team has generated transgenic rabbit and mouse models of HCM and shown that cardiac hypertrophy and fibrosis could be reversed through genetic or pharmacological interventions. Results with NAC, a precursor to glutathione, the largest intracellular thiol pool against oxidative stress, were most promising. In three independent studies in two different transgenic models of HCM (rabbits and mouse), treatment with NAC completely reversed cardiac hypertrophy and fibrosis and improved indices of diastolic function. The ultimate goal of every physician-scientist is to apply the bench discoveries at the bedside. The study team proposes to test their findings in the animal models in humans with HCM caused by sarcomere protein mutations. The use of NAC is also supported by data showing increased oxidative stress in human HCM. Moreover, NAC has been used extensively in humans and has a well-established safety profile. Resources including patients with sarcomere protein mutations are available to successfully complete a randomized placebo-controlled (N=25) pilot study to test two escalating doses of NAC (N=50), administered for one year. The study aims to determine recruitment, accrual, retention and compliance rates; tolerability, safety and side effects; and estimate the effect size of NAC on the indices of cardiac hypertrophy at the baseline and after one year of treatment. Only HCM patients with sarcomere proteins mutations will be included to exclude phenocopy. The Core centers will interpret the phenotypic data to assure homogeneity. Data Coordinating Center will assist in the research design, planning and conduct of the study and analysis of the data. The findings will set the stage for large-scale robust randomized placebo-control efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary cardiac hypertrophy, non-dilated LV cavity and preserved LV systolic function, hence, the diagnosis of HCM, who have at least an LV end diastolic (LVSD) wall thickness of at least 15 mm on a 2D echocardiogram and
* Known to have mutations in genes encoding sarcomeric proteins

Exclusion Criteria:

* Hypersensitivity to NAC
* Individuals younger than 18 years old (in the pilot study)
* Phenocopy conditions, diagnosed clinically or genetically
* Patients who have undergone transcatheter (alcohol) septal ablation within 6 months.
* Individuals (typically family members) with causal mutations but an LVSD wall thickness of <15 mm
* Patients with concomitant diseases such as:

  * Significant coronary artery disease >70% luminal diameter stenosis in ny of the major coronary arteries (if known);
  * Valvular heart diseases (more than mild aortic stenosis and mitral regurgitation, the latter judged to be due to primary mitral valve abnormalities);
  * Uncontrolled hypertension, defined as systolic blood pressure of

    * 140 mmHg and diastolic blood pressure of ≥90 mmHg on medication, mean of three measurements at rest);
  * Other significant medical problems, such as moderate to severe chronic renal failure (GFR<45 ml/min/1.73m2), advanced liver disease, cancer, or other disabling conditions
* Pregnant women, nursing mothers and those who plan pregnancy during the study period
* Those with active asthma (albeit the concern is relevant to nebulizer form but not oral formulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali J. Marian, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Marian AJ, Tan Y, Li L, Chang J, Syrris P, Hessabi M, Rahbar MH, Willerson JT, Cheong BY, Liu CY, Kleiman NS, Bluemke DA, Nagueh SF. Hypertrophy Regression With N-Acetylcysteine in Hypertrophic Cardiomyopathy (HALT-HCM): A Randomized, Placebo-Controlled, Double-Blind Pilot Study. Circ Res. 2018 Apr 13;122(8):1109-1118. doi: 10.1161/CIRCRESAHA.117.312647. Epub 2018 Mar 14. PMID 29540445

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine (NAC): N-acetylcysteine (NAC) 600mg by mouth every 12 hours for 90 days. N-acetylcysteine 1200mg by mouth every 12 hours for 270 days
  N-acetylcysteine: NAC 600mg capsule or matching Placebo , 1 twice daily for 90 days, then increase to NAC 1,200mg or matching placebo, 2 capsules twice daily for 270 days.
Period: Overall Study
Arm/Group | N-acetylcysteine (NAC) | Placebo
Started | 29 | 13
Completed | 24 | 11
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine (NAC) | Placebo | Total
Number analyzed (Participants) | 29 | 13 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 34
  >=65 years | 7 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.0) | 47.6 (15.1) | 49.15 (0.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 22 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 25 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Recruitment as Assessed by Number of Participants Who Enrolled to the Study
Time Frame: at the time of enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo 1 cap by mouth every 12 hours for 90 days. Placebo 2 caps by mouth every 12 hours for 270 days.
  Placebo: sugar pill manufactured to mimic NAC 600mg capsule
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 29 | 13
Participants | 29 | 13

2. Primary Outcome: Retention as Assessed by Number of Participants Who Completed the Study
Time Frame: from baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 29 | 13
Participants | 24 | 11

3. Primary Outcome: Compliance as Assessed by Percentage of Pills Taken by Participant
Description: Participants returned all pill bottles to the study team, and the number of pills not taken by the participant (that is, the number of pills remaining in the bottles) were counted. Compliance is reported as percentage of pills taken by the participant.
Time Frame: from baseline to 12 months
Population: Data are reported for participants for whom all pill bottles were returned to the study team. It was not known whether the returned bottles contained placebo or NAC; therefore, the data for both arms are reported together.
Measure: Mean (Standard Deviation); unit: percentage of pills taken
Groups:
- All Participants: N-acetylcysteine: NAC 600mg capsule or matching Placebo , 1 twice daily for 90 days, then increase to NAC 1,200mg or matching placebo, 2 capsules twice daily for 270 days.
  OR
  Placebo: sugar pill manufactured to mimic NAC 600mg capsule
Arm/Group | All Participants
Number analyzed (Participants) | 30
percentage of pills taken | 92 (0.0878)

4. Primary Outcome: Number of Participants With Side Effects Attributable to the Intervention
Time Frame: from baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 29 | 13
Participants | 0 | 0

5. Primary Outcome: Interventricular Septal Thickness (IVST) as Assessed by Echocardiography
Time Frame: baseline
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
millimeters (mm) | 18.88 (4.59) | 18.00 (3.97)

6. Primary Outcome: Interventricular Septal Thickness (IVST) as Assessed by Echocardiography
Time Frame: 12 months
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
millimeters (mm) | 17.92 (3.3) | 17.82 (4.87)

7. Secondary Outcome: Left Ventricular End-systolic Diameter (LVESD) as Assessed by Echocardiography
Time Frame: 12 months
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
millimeters (mm) | 21.88 (5.29) | 21.55 (3.8)

8. Secondary Outcome: Left Ventricular End-systolic Diameter (LVESD) as Assessed by Echocardiography
Time Frame: baseline
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
millimeters (mm) | 22.13 (6.06) | 22.64 (5.16)

9. Secondary Outcome: Left Ventricular Mass (LVM) as Assessed by Echocardiography
Description: Left Ventricular Mass (LVM) is the weight of the left heart and is estimated from the echocardiographic measurements that include left ventricular wall thickness and the chamber diameter. The weight is calculated in grams and then normalized to body surface area (m^2), with LVM reported as g/m^2.
Time Frame: baseline
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
g/m^2 | 269.65 (94.17) | 292.80 (107.50)

10. Secondary Outcome: Left Ventricular Mass (LVM) as Assessed by Echocardiography
Description: as for outcome 9
Time Frame: 12 months
Population: Data are reported for all participants who completed the study.
Measure: Mean (Standard Deviation); unit: g/m^2
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 24 | 11
g/m^2 | 281.98 (81.75) | 290.44 (99.81)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Placebo: Placebo 1 cap by mouth every 12 hours for 90 days. Placebo 2 caps by mouth every 12 hours for 270 days.
  N-acetylcysteine: NAC 600mg capsule or matching Placebo , 1 twice daily for 90 days, then increase to NAC 1,200mg or matching placebo, 2 capsules twice daily for 270 days.
  Placebo: sugar pill manufactured to mimic NAC 600mg capsule
Arm/Group | N-acetylcysteine (NAC) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/13
Serious Adverse Events (participants affected / at risk) | 5/29 | 0/13
Other Adverse Events (participants affected / at risk) | 2/29 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (NAC) (N=29) | Placebo (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Event was not related to administration of NAC.
Cerebrovascular accident (Vascular disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (NAC) (N=29) | Placebo (N=13)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 — Event is not related to NAC.

LIMITATIONS AND CAVEATS:
The small sample size of the study prohibits from making firm conclusions about efficacy of NAC in hypertrophic cardiomyopathy (HCM).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No